CLINICAL TRIAL: NCT00023712
Title: A Phase II Evaluation of Bortezomib (Velcade™, PS-341, NSC #681239, IND #58443) in the Treatment of Persistent or Recurrent Platinum-Sensitive Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: Bortezomib in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02404; NCI-2012-02404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068853; GOG-0146N; GOG #0146N (Other: Gynecologic Oncology Group); GOG-0146N (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of bortezomib in treating patients who have persistent or recurrent ovarian epithelial cancer or primary peritoneal cancer. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of bortezomib in patients with persistent or recurrent platinum-sensitive ovarian epithelial or primary peritoneal carcinoma.

II. Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent or recurrent ovarian epithelial or primary peritoneal carcinoma
* Measurable disease

  * At least 20 mm by conventional techniques (e.g., palpation, x-ray, plain CT scan, or MRI) OR at least 10 mm by spiral CT scan
* Must have had prior therapy with no more than 1 platinum-based chemotherapy regimen for primary disease (e.g., carboplatin, cisplatin, or other organoplatinum compound)

  * A second regimen containing paclitaxel allowed provided patient received no prior paclitaxel therapy
* Platinum-sensitive disease

  * Treatment-free interval without progressive disease for more than 6 months but less than 12 months after therapy with platinum-based regimen
* At least 1 target lesion outside previously irradiated field
* Ineligible for higher priority GOG protocol
* Performance status - GOG 0-2 (if received 1 prior therapy regimen)
* Performance status - GOG 0-1 (if received 2 prior therapy regimens)
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No evidence of acute ischemia or significant conduction abnormality (e.g., left anterior hemiblock in the presence of right bundle branch block or second or third degree atrioventricular block) on electrocardiogram
* No myocardial infarction within the past 6 months
* No cerebrovascular event or transient ischemic attack within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except non-melanoma skin cancer
* No sensory or motor neuropathy greater than grade 1
* No more than 1 prior non-cytotoxic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule inhibitors of signal transduction) for recurrent or persistent disease
* At least 4 weeks since prior biological or immunological agents and recovered
* No prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimen
* At least 4 weeks since prior chemotherapy and recovered
* At least 1 week since prior anti-cancer hormonal therapy and recovered
* Concurrent hormone replacement therapy allowed
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to target lesions
* No prior radiotherapy to more than 25% of marrow-bearing areas
* At least 4 weeks since prior surgery and recovered
* No prior bortezomib
* No prior anti-cancer therapy that would preclude study treatment
* No concurrent amifostine or other protective agents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2001-11-05 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual was broken down into two cohorts. Cohort 1 enrolled 28 participants from 11/5/2001 through 1/6/2003. Cohort 2 enrolled 30 participants from 4/5/2004 through 9/6/2005.
Groups:
- Cohort 1 - Bortezomib (1.5 mg/m2): Patients enrolled 11/5/2001 through 1/6/2003 receive bortezomib 1.5 mg/m2/dose IV twice weekly for 2 weeks (Days 1,4,8, and 11) followed by a 10day rest period (Days 12-21). At least 72 hours should elapse between consecutive doses.Courses repeat every 3 weeks (21 days) until disease progression or adverse effects prohibit further therapy.
- Cohort 2 - Bortezomib (1.3 mg/m2): Patients enrolled 4/5/2004 through 9/6/2005 receive bortezomib 1.3 mg/m2/dose IV twice weekly for 2 weeks (Days 1,4,8, and 11) followed by a 10day rest period (Days 12-21). At least 72 hours should elapse between consecutive doses.Courses repeat every 3 weeks (21 days) until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Cohort 1 - Bortezomib (1.5 mg/m2) | Cohort 2 - Bortezomib (1.3 mg/m2)
Started | 28 (total number of participants enrolled on study) | 30 (total number of participants enrolled on study)
Completed | 26 (total number of participants eligible and evaluable) | 29 (total number of participants eligible and evaluable)
Not Completed | 2 | 1
Not completed — Not platinum sensitive | 1 | 0
Not completed — Never treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Cohort 1: 2 participants were not eligible/evaluable after enrollment. Cohort 2: 1 participant was not eligible/evaluable after enrollment.
Groups:
- Cohort 1: Patients enrolled 11/5/2001 through 1/6/2003 receive bortezomib 1.5 mg/m2/dose IV twice weekly for 2 weeks (Days 1,4,8, and 11) followed by a 10day rest period (Days 12-21). At least 72 hours should elapse between consecutive doses.Courses repeat every 3 weeks (21 days) until disease progression or adverse effects prohibit further therapy.
- Cohort 2: Patients enrolled 4/5/2004 through 9/6/2005 receive bortezomib 1.3 mg/m2/dose IV twice weekly for 2 weeks (Days 1,4,8, and 11) followed by a 10day rest period (Days 12-21). At least 72 hours should elapse between consecutive doses.Courses repeat every 3 weeks (21 days) until disease progression or adverse effects prohibit further therapy.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.1) | 55.8 (11.4) | 57.2 (11.2)
Age, Customized [Number; unit: participants]
  20-29 years | 0 | 1 | 1
  30-39 years | 1 | 1 | 2
  40-49 years | 6 | 4 | 10
  50-59 years | 8 | 10 | 18
  60-69 years | 6 | 11 | 17
  70-79 years | 5 | 1 | 6
  80-89 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 3
  United States | 23 | 29 | 52
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1 | 0 | 1
  Endometrioid Adenocarcinoma | 1 | 1 | 2
  Mixed Epithelial Carcinoma | 2 | 1 | 3
  Serous Adenocarcinoma | 21 | 25 | 46
  Transitional Cell Carcinoma | 1 | 1 | 2
  Undifferentiated Carcinoma | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Duration
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: From study entry, up to 5 years
Measure: Median (Full Range); unit: months
Groups:
- Cohort 1 - Bortezomib 1.5 (mg/m2): Patients enrolled 11/5/2001 through 1/6/2003 receive bortezomib 1.5 mg/m2/dose IV twice weekly for 2 weeks (Days 1,4,8, and 11) followed by a 10day rest period (Days 12-21). At least 72 hours should elapse between consecutive doses.Courses repeat every 3 weeks (21 days) until disease progression or adverse effects prohibit further therapy.
Arm/Group | Cohort 1 - Bortezomib 1.5 (mg/m2) | Cohort 2 - Bortezomib (1.3 mg/m2)
Number analyzed (Participants) | 26 | 29
months | 3.9 [3.9 to 3.9] | 24.1 [2.4 to 45.9]

2. Primary Outcome: Frequency and Severity of Observed Adverse Events
Time Frame: Up to 5 years
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0 AEs Cohort 1 - Bortezomib 1.5 (mg/m2): Number of patients who did not experience the specified AE in cohort 1.
- Grade 1 AEs (CTCAE v.2.0) Cohort 1 - Bortezomib 1.5 (mg/m2): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 2.0 in cohort 1
- Grade 2 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 2.0 in Cohort 1.
- Grade 3 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 2.0 in cohort 1
- Grade 4 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 2.0 in cohort 1.
- Grade 0 AEs Cohort 2 - Bortezomib (1.3 mg/m2): Number of patients who did not experience the specified AE in cohort 2
- Grade 1 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 2.0 in cohort 2.
- Grade 2 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 2.0 in cohort 2
- Grade 3 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 2.0 in cohort 2.
- Grade 4 AEs (CTCAE v 2.0) Cohort 2- Bortezomib (1.3 mg/m2): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 2.0 in cohort 2.
Arm/Group | Grade 0 AEs Cohort 1 - Bortezomib 1.5 (mg/m2) | Grade 1 AEs (CTCAE v.2.0) Cohort 1 - Bortezomib 1.5 (mg/m2) | Grade 2 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2) | Grade 3 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2) | Grade 4 AEs (CTCAE v 2.0) Cohort 1 - Bortezomib 1.5 (mg/m2) | Grade 0 AEs Cohort 2 - Bortezomib (1.3 mg/m2) | Grade 1 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2) | Grade 2 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2) | Grade 3 AEs (CTCAE v 2.0) Cohort 2 - Bortezomib (1.3 mg/m2) | Grade 4 AEs (CTCAE v 2.0) Cohort 2- Bortezomib (1.3 mg/m2)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 29 | 29 | 29 | 29 | 29
Participants
  Platelets | 14 | 9 | 0 | 3 | 0 | 16 | 10 | 3 | 0 | 0
  Absolute neutrophil count (ANC) | 18 | 5 | 2 | 1 | 0 | 21 | 5 | 3 | 0 | 0
  Fatigue | 4 | 10 | 10 | 1 | 1 | 7 | 11 | 6 | 5 | 0
  Rash | 14 | 6 | 4 | 2 | 0 | 17 | 9 | 3 | 0 | 0
  Diarrhea | 13 | 7 | 2 | 4 | 0 | 21 | 5 | 3 | 0 | 0
  Constipation | 17 | 4 | 5 | 0 | 0 | 11 | 7 | 9 | 0 | 2
  Genitourinary/renal | 24 | 1 | 0 | 1 | 0 | 25 | 3 | 1 | 0 | 0
  Hepatic | 21 | 3 | 1 | 0 | 1 | 22 | 6 | 1 | 0 | 0
  Infection | 23 | 1 | 1 | 0 | 1 | 25 | 2 | 2 | 0 | 0
  Metabolic | 21 | 3 | 0 | 2 | 0 | 24 | 4 | 1 | 0 | 0
  Neuropathy (sensory) | 14 | 6 | 3 | 3 | 0 | 15 | 8 | 4 | 2 | 0
  Pain | 12 | 8 | 5 | 1 | 0 | 15 | 5 | 7 | 2 | 0
  Pulmonary | 21 | 0 | 3 | 2 | 0 | 26 | 0 | 2 | 1 | 0

3. Primary Outcome: Objective Partial/Complete Tumor Response Based on the Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Number of participants who experienced an objective tumor response up to 5 years. Per RECIST version 1.0 criteria: each target lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or >= 10 mm when measured by spiral CT. Complete Response is a disappearance of all target and non-target lesions. Partial Response is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions, taking as reference the baseline sum of LD.
Time Frame: From study entry until disease progression/intolerable toxicity/study withdrawal
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Bortezomib 1.5 (mg/m2) | Cohort 2 - Bortezomib (1.3 mg/m2)
Number analyzed (Participants) | 26 | 29
participants | 1 | 2

4. Secondary Outcome: Overall Survival
Time Frame: From study entry, up to 5 years following disease progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Bortezomib 1.5 (mg/m2) | Cohort 2 - Bortezomib (1.3 mg/m2)
Number analyzed (Participants) | 26 | 29
months | 18.2 [13.0 to 29.0] | 27.2 [12.7 to 37.1]

5. Secondary Outcome: Progression-Free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: From study entry up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Bortezomib 1.5 (mg/m2) | Cohort 2 - Bortezomib (1.3 mg/m2)
Number analyzed (Participants) | 26 | 29
months | 1.5 [1.3 to 4.8] | 1.4 [1.4 to 3.1]

ADVERSE EVENTS:
Time Frame: All Adverse Events(AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 5/26 | 6/29
Other Adverse Events (participants affected / at risk) | 26/26 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=26) | Cohort 2 (N=29)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Caridic Left Ventricular Function (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Gi Other (Gastrointestinal disorders) | 0 | 1
Sgot(Ast) (Hepatobiliary disorders) | 1 | 0
Cns Cerebrovascular Ischemia (Nervous system disorders) | 0 | 1
Neuropathic Pain (General disorders) | 1 | 0
Headache (General disorders) | 0 | 1
Myalgia (General disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=26) | Cohort 2 (N=29)
Inner Ear/Hearing (Ear and labyrinth disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 14
Leukopenia (Blood and lymphatic system disorders) | 6 | 9
Transfusion Prbc's (Blood and lymphatic system disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 18 | 17
Edema (Cardiac disorders) | 3 | 1
Fever(No Neutropenia) (General disorders) | 3 | 5
Weight Gain(No Vod) (General disorders) | 2 | 1
Fatigue (General disorders) | 21 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Rash Desquamation (Skin and subcutaneous tissue disorders) | 10 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Anorexia (Gastrointestinal disorders) | 5 | 8
Diarrhea Without Colostomy (Gastrointestinal disorders) | 11 | 8
Constipation (Gastrointestinal disorders) | 10 | 18
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 4 | 3
Vomitting (Gastrointestinal disorders) | 8 | 10
Nausea (Gastrointestinal disorders) | 15 | 13
Gi Other (Gastrointestinal disorders) | 2 | 0
Hypoalbuminemia (Hepatobiliary disorders) | 1 | 3
Sgot(Alt) (Hepatobiliary disorders) | 4 | 7
Sgot(Ast) (Hepatobiliary disorders) | 1 | 4
Alkaline Phosphatase (Hepatobiliary disorders) | 2 | 3
Infection Without Neutropenia (Infections and infestations) | 3 | 7
Metabolic Other (Metabolism and nutrition disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 6
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Confusion (Nervous system disorders) | 2 | 1
Mood Alteration Anxiety/Agitation (Nervous system disorders) | 1 | 5
Insomnia (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 1 | 3
Mood Alteration Depression (Nervous system disorders) | 3 | 7
Neuropathy Sensor (Nervous system disorders) | 11 | 14
Ocular Other (Eye disorders) | 0 | 3
Vision Flashing Lights/Floaters (Eye disorders) | 2 | 0
Vision Blurres (Eye disorders) | 1 | 3
Abdominal Pain (General disorders) | 11 | 13
Pain Other (General disorders) | 6 | 7
Neuropathic Pain (General disorders) | 0 | 4
Headache (General disorders) | 5 | 9
Chest Pain (General disorders) | 3 | 1
Bone Pain (General disorders) | 1 | 4
Arthralgia (General disorders) | 5 | 6
Myalgia (General disorders) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Creatinine (Renal and urinary disorders) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less